CLINICAL TRIAL: NCT02298842
Title: In Vitro Study of Platelets Collected on Trima Accel System and Stored in InterSol Solution
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Terumo BCT (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: CTS-5051
Record Dates: First submitted 2014-11-14; First posted 2014-11-24 (Estimated); Results first posted 2017-07-14 (Actual); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Healthy Volunteers
Keywords: Healthy Adults

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Platelets Stored in Plasma (Active Comparator): Platelets stored in Plasma
  Interventions: Device: Platelets stored in Plasma
- Test Platelets Stored in InterSol (Experimental): Platelets stored in InterSol
  Interventions: Device: Platelets stored in InterSol

INTERVENTIONS:
Device: Platelets stored in InterSol — A platelet apheresis procedure involves connecting the blood in the donor's vein through tubing to a machine that separates the blood components. After the separation, the desired component of the blood is removed (platelets and plasma), while the remainder of the blood components are reinfused back into the patient. To prevent clotting, an anticoagulant (ACDA) is used throughout the procedure. Following each blood collection, Platelet Additive Solution (PAS), InterSol, will be added to the platelet product to prepare the final product for 7 day storage. The entire procedure is painless and should take 90 to 120 minutes and the subjects will have two collections within 6-8 days of each other.
  Arms: Test Platelets Stored in InterSol
Device: Platelets stored in Plasma — A platelet apheresis procedure involves connecting the blood in the donor's vein through tubing to a machine that separates the blood components. After the separation, the desired component of the blood is removed (platelets and plasma), while the remainder of the blood components are reinfused back into the patient. To prevent clotting, an anticoagulant (ACDA) is used throughout the procedure. During the collection, plasma collected from the donor will be added to the platelet product to prepare the final product for 7 day storage. The entire procedure is painless and should take 90 to 120 minutes and the subjects will have two collections within 6-8 days of each other.
  Arms: Platelets Stored in Plasma

SUMMARY:
This study sought to verify that the in vitro quality (functional assays) of platelets collected on the Trima Accel system, Version 6.4, diluted in InterSol Solution, and stored for 1, 5, and 7 days meet FDA requirements.

DETAILED DESCRIPTION:
Platelets suspended in platelet additive solutions (PAS) have been collected and transfused in Europe for over 20 years. These PAS solutions outside of the United States (US) are not tied to an apheresis device; however in the US, PAS solutions have traditionally been linked to a corresponding apheresis device.

Currently in the US, there are two solutions approved by the Food and Drug Administration (FDA) as a PAS for the replacement of 65% plasma in platelet components. Isoplate Solution is approved for use with the Trima Accel® Automated Blood Collection System (Trima Accel System) and InterSol Solution is approved for use with the Amicus Separator System.

This study is designed to provide blood centers with the option to use either Isoplate or InterSol when collecting platelets for use with PAS. Terumo BCT is pursuing approval for InterSol Solution in combination with the Trima Accel System.

This is a randomized, paired, prospective, open-label, multi-center study. Up to 120 healthy adult subjects will be enrolled in this study to ensure 60 paired evaluable data points across two Investigational Sites. Evaluable is defined as two completed platelet products with 100mL plasma that do not meet any of the protocol analysis exclusion criteria.

The additional platelet donors account for screen failures, incomplete procedures, and protocol exclusions.

Two units of platelets will be collected from each subject: one Test unit collected as a hyperconcentrated platelet product with 100 mL of concurrent plasma and one Control unit of platelets in plasma collected according to standard procedure. The Test unit will be suspended in 65% Intersol/35% plasma immediately after collection; the Control unit will be maintained in 100% plasma.

Eligible donors who have signed an informed consent will be enrolled. Randomization will occur in a ratio of 1:1 to one of the following Treatment Arms:

Arm A: Collection of one Test unit followed by collection of one Control unit Arm B: Collection of one Control unit followed by collection of one Test unit

The standard apheresis platelet units collected in the Control arm will mirror the hyperconcentrated platelet units in the Test arm in terms of yield and final concentration.

SUBJECT PROCEDURES

Screening can be performed within 30 days of the apheresis procedure or combined with the first Apheresis Visit.

The following evaluations will be performed:

1. Informed consent will be obtained prior to initiating any study specific procedures
2. Eligibility will be confirmed
3. Demographics (age, gender, ethnic origin), height, and weight
4. Complete blood count (CBC) for hemoglobin and platelet count on subjects new to the Investigative Site that do not have historical hemoglobin and/or platelet count measurements

Apheresis Visit

The following procedures will be performed at both the first and second Apheresis Visits:

1. Eligibility will be confirmed
2. Finger stick hemoglobin
3. First apheresis procedure will be performed

Subject will return to the Site in 6 to 8 days following the first apheresis collection for the second apheresis collection. This will conclude the subject's participation.

Apheresis procedures will be run according to the instructions and precautions described in the commercially available Trima Accel Operator's Manual for use with Version 6.4.

The Investigator or designee will perform the venipuncture, monitor the subject during the collection, assess and provide any interventions for adverse effects, remove the needle, dress the puncture site and monitor subject through recovery.

The following will be documented:

1. Trima Procedure details
2. Adverse events
3. Medications to treat AEs
4. Device deficiencies

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years of age or older
* Meet the inclusion criteria defined by the Investigational Site for an apheresis double platelet with plasma collection on the Trima Accel System. These criteria are based on American Association of Blood Banks (AABB) standards. Note: Subjects who are deferred from volunteer community donations because of travel restrictions, piercings or tattoos may participate in the study.

Exclusion Criteria:

* None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2015-11-05; Primary Completion 2016-05-12 (Actual); Study Completion 2016-05-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jose Cancelas-Perez, MD, PhD, Principal Investigator — Hoxworth Blood Center; Mehraboon S Irani, MD, Principal Investigator — Clood Center of Wisconsin
Locations (2):
- United States (2):
  - Hoxworth Blood Center, Cincinnati, Ohio
  - Blood Center of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dumont LJ, Cancelas JA, Graminske S, Friedman KD, Vassallo RR, Whitley PH, Rugg N, Dumont DF, Herschel L, Siegal AH, Szczepiorkowski ZM, Fender L, Razatos A. In vitro and in vivo quality of leukoreduced apheresis platelets stored in a new platelet additive solution. Transfusion. 2013 May;53(5):972-80. doi: 10.1111/j.1537-2995.2012.03841.x. Epub 2012 Aug 6. PMID 22882530
- [Background] Ringwald J, Walz S, Zimmermann R, Zingsem J, Strasser E, Weisbach V, Eckstein R. Hyperconcentrated platelets stored in additive solution: aspects on productivity and in vitro quality. Vox Sang. 2005 Jul;89(1):11-8. doi: 10.1111/j.1423-0410.2005.00645.x. PMID 15938735
- [Background] Cohn CS, Stubbs J, Schwartz J, Francis R, Goss C, Cushing M, Shaz B, Mair D, Brantigan B, Heaton WA. A comparison of adverse reaction rates for PAS C versus plasma platelet units. Transfusion. 2014 Aug;54(8):1927-34. doi: 10.1111/trf.12597. Epub 2014 Apr 16. PMID 24735171
- [Background] Diedrich B, Sandgren P, Jansson B, Gulliksson H, Svensson L, Shanwell A. In vitro and in vivo effects of potassium and magnesium on storage up to 7 days of apheresis platelet concentrates in platelet additive solution. Vox Sang. 2008 Feb;94(2):96-102. doi: 10.1111/j.1423-0410.2007.01002.x. Epub 2007 Nov 22. PMID 18034788
- [Background] Gulliksson H, AuBuchon JP, Vesterinen M, Sandgren P, Larsson S, Pickard CA, Herschel I, Roger J, Tracy JE, Langweiler M; Biomedical Excellence for Safer Transfusion Working Party of the International Society of Blood Transfusion. Storage of platelets in additive solutions: a pilot in vitro study of the effects of potassium and magnesium. Vox Sang. 2002 Apr;82(3):131-6. doi: 10.1046/j.1423-0410.2002.drfgv158.x. PMID 11952987
- [Background] Dumont LJ, VandenBroeke T, Ault KA. Platelet surface P-selectin measurements in platelet preparations: an international collaborative study. Biomedical Excellence for Safer Transfusion (BEST) Working Party of the International Society of Blood Transfusion (ISBT). Transfus Med Rev. 1999 Jan;13(1):31-42. doi: 10.1016/s0887-7963(99)80086-8. No abstract available. PMID 9924762

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 87 volunteers signed consent and were enrolled in the study, but 2 were screen fails and therefore did not participate in the study
Groups:
- InterSol First, Then Plasma: Platelets collected in InterSol, then platelets collected in plasma
- Plasma First, Then InterSol: Platelets collected in plasma, then platelets collected in InterSol
Period: First Platelet Donation (Day 0)
Arm/Group | InterSol First, Then Plasma | Plasma First, Then InterSol
Started | 44 | 41
Completed | 38 | 36
Not Completed | 6 | 5
Period: Second Platelet Donation (Day 6-8)
Arm/Group | InterSol First, Then Plasma | Plasma First, Then InterSol
Started | 38 | 36
Completed | 30 | 30
Not Completed | 8 | 6

BASELINE CHARACTERISTICS:
Population: The Safety Population includes all participants enrolled in this study who underwent any study related apheresis procedure.
Groups:
- Total: Total of all reporting groups
Arm/Group | InterSol First, Then Plasma | Plasma First, Then InterSol | Total
Number analyzed (Participants) | 44 | 41 | 85
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 41 | 37 | 78
  >=65 years | 3 | 4 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.9 (14.10) | 43.3 (14.98) | 42.1 (14.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 13 | 28
  Male | 29 | 28 | 57
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 43 | 40 | 83
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 44 | 41 | 85
Height [Mean (Standard Deviation); unit: inches] | 69.5 (3.12) | 68.5 (3.43) | 69.0 (3.30)
Weight [Mean (Standard Deviation); unit: lbs] | 197.9 (34.38) | 188.7 (30.87) | 193.4 (32.87)
Total Blood Volume (TBV) [Mean (Standard Deviation); unit: mL] | 5380.1 (770.93) | 5172.5 (757.45) | 5280.0 (767.04)

OUTCOME MEASURES:

1. Primary Outcome: pH of Platelets at Day 5
Description: The primary endpoint for this study is pH of platelets stored in InterSol at Day 5. The FDA acceptance criteria for pH is 95% of products have pH >6.2 at 22 degrees C with 95% confidence interval. A sample size of 60 subjects was chosen for the study to meet the acceptance criteria with 0 failures out of 60 Test products.
Time Frame: Day 5
Population: The Full Analysis Set (FAS) was used to examine the primary and secondary endpoints.The FAS consisted of all products where the corresponding Test and Control values for the primary endpoint did not meet any of the protocol analysis exclusion criteria.
Measure: Mean (Standard Deviation); unit: pH
Groups:
- Test Platelets Collected and Stored in InterSol: Platelets stored in InterSol
  Platelets stored in InterSol: A platelet apheresis procedure involves connecting the blood in the donor's vein through tubing to a machine that separates the blood components. After the separation, the desired component of the blood is removed (platelets and plasma), while the remainder of the blood components are reinfused back into the patient. To prevent clotting, an anticoagulant (ACDA) is used throughout the procedure. Following each blood collection, Platelet Additive Solution (PAS), InterSol, will be added to the platelet product to prepare the final product for 7 day storage. The entire procedure is painless and should take 90 to 120 minutes and the subjects will have two collections within 6-8 days of each other.
- Control Platelets Collected and Stored in Plasma: Platelets stored in Plasma
  Platelets stored in Plasma: A platelet apheresis procedure involves connecting the blood in the donor's vein through tubing to a machine that separates the blood components. After the separation, the desired component of the blood is removed (platelets and plasma), while the remainder of the blood components are reinfused back into the patient. To prevent clotting, an anticoagulant (ACDA) is used throughout the procedure. During the collection, plasma collected from the donor will be added to the platelet product to prepare the final product for 7 day storage. The entire procedure is painless and should take 90 to 120 minutes and the subjects will have two collections within 6-8 days of each other.
Arm/Group | Test Platelets Collected and Stored in InterSol | Control Platelets Collected and Stored in Plasma
Number analyzed (Participants) | 60 | 60
pH | 7.184 (0.0718) | 7.414 (0.0975)
Statistical Analysis 1: Comparison: Test Platelets Collected and Stored in InterSol vs Control Platelets Collected and Stored in Plasma; A "success" is defined as pH22°C at Day 5 and Day 7 being at least 6.2. A one-sided 95% lower confidence limit will be used to assess the proportion of successes at Day 5 and Day 7. If the lower limit of the one-sided 95% confidence interval exceeds 0.95, the Test product will meet the FDA acceptance criteria; Test type: Non-Inferiority — The sample size of 60 was chosen to meet the FDA pH requirements that the lower 95% confidence limit on the proportion of platelet test units with pH> 6.2 will be at least 95%. This will be achieved if zero failures (pH<=6.2) is seen; Exact Binomial Confidence Interval; Simple sample proportion = 100, 95% CI 1-sided [lower limit 95.1], Standard Deviation 0 — Estimated proportion is 100%. Hence standard deviation is estimated as 0

2. Primary Outcome: pH of Platelets at Day 7
Description: The primary endpoint for this study is pH of platelets stored in InterSol at Day 7. The FDA acceptance criteria for pH is 95% of products have pH >6.2 at 22 degrees C with 95% confidence interval. A sample size of 60 subjects was chosen for the study to meet the acceptance criteria with 0 failures out of 60 Test products.
Time Frame: Day 7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Test Platelets Collected and Stored in InterSol | Control Platelets Collected and Stored in Plasma
Number analyzed (Participants) | 60 | 60
pH | 7.152 (0.0855) | 7.335 (0.1313)
Statistical Analysis 1: Comparison: Test Platelets Collected and Stored in InterSol vs Control Platelets Collected and Stored in Plasma; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Exact Bionomial Confidence Interval; Simple sample proportion = 100, 95% CI 1-sided [lower limit 95.1], Standard Deviation 0 — Estimated proportion is 100%. Hence standard deviation is estimated as 0

3. Secondary Outcome: Percent of Platelets Activated as Measured by P-selectin
Description: Flow cytometric detection of platelet P-selectin expression (Units: %). Lower value is considered to indicate better platelet quality.
Time Frame: Day 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent of Platelets Activated
Arm/Group | Test Platelets Collected and Stored in InterSol | Control Platelets Collected and Stored in Plasma
Number analyzed (Participants) | 60 | 60
Percent of Platelets Activated | 26.324 (7.6052) | 9.354 (4.4110)
Statistical Analysis 1: Comparison: Test Platelets Collected and Stored in InterSol vs Control Platelets Collected and Stored in Plasma; The null hypothesis is that P-selectin's mean difference, Test - 1.25 * Control, is greater than or equal to 0, and the alternative is that the mean difference is less than 0; Test type: Non-Inferiority — If the 97.5% upper limit of the confidence interval is less than 0, the null hypothesis will be rejected in favor of the alternative suggesting the Test product is not inferior to the Control product; Mean Difference (Final Values) = 15.099, 97.5% CI 1-sided [upper limit 16.738], Standard Deviation 5.6367 — Estimated from an ANCOVA with effects of treatment and subject nested within sequence

4. Secondary Outcome: Percent of Extent of Shape Change
Description: Measures the proportion of platelets that have a discoid morphology (Units: %). Higher value is considered to indicate better platelet quality.
Time Frame: Day 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: % extent of shape change
Groups:
- Arm A - Test Platelets Stored in InterSol: Platelets stored in InterSol
  Platelets stored in InterSol: A platelet apheresis procedure involves connecting the blood in the donor's vein through tubing to a machine that separates the blood components. After the separation, the desired component of the blood is removed (platelets and plasma), while the remainder of the blood components are reinfused back into the patient. To prevent clotting, an anticoagulant (ACDA) is used throughout the procedure. Following each blood collection, Platelet Additive Solution (PAS), InterSol, will be added to the platelet product to prepare the final product for 7 day storage. The entire procedure is painless and should take 90 to 120 minutes and the subjects will have two collections within 6-8 days of each other.
- Arm B - Platelets Stored in Plasma: Platelets stored in Plasma
  Platelets stored in Plasma: A platelet apheresis procedure involves connecting the blood in the donor's vein through tubing to a machine that separates the blood components. After the separation, the desired component of the blood is removed (platelets and plasma), while the remainder of the blood components are reinfused back into the patient. To prevent clotting, an anticoagulant (ACDA) is used throughout the procedure. During the collection, plasma collected from the donor will be added to the platelet product to prepare the final product for 7 day storage. The entire procedure is painless and should take 90 to 120 minutes and the subjects will have two collections within 6-8 days of each other.
Arm/Group | Arm A - Test Platelets Stored in InterSol | Arm B - Platelets Stored in Plasma
Number analyzed (Participants) | 60 | 60
% extent of shape change | 24.109 (5.9968) | 30.658 (5.1498)
Statistical Analysis 1: Comparison: Arm A - Test Platelets Stored in InterSol vs Arm B - Platelets Stored in Plasma; The null hypothesis is that ESC's mean difference, Test - 0.8 * Control, is less than or equal to 0, and the alternative is that the mean difference is greater than 0; Test type: Non-Inferiority — Higher value is considered to indicate better platelet quality. If the 97.5% lower limit of the confidence interval is greater than 0, the null hypothesis will be rejected in favor of the alternative suggesting the Test product is not inferior to the Control product; Median Difference (Final Values) = -0.418, 97.5% CI 1-sided [lower limit -1.544], Standard Deviation 4.5531 — Estimated from an ANCOVA with effects of treatment and subject nested within sequence

5. Secondary Outcome: Percent of Platelets Exhibiting Hypotonic Shock Response
Description: Measures the ability of platelets to recover their volume after being exposed to a hypotonic environment (Units: % Recovery). Higher value is considered to indicate better platelet quality.
Time Frame: Day 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: % of hypotonic shock response
Arm/Group | Test Platelets Collected and Stored in InterSol | Control Platelets Collected and Stored in Plasma
Number analyzed (Participants) | 60 | 60
% of hypotonic shock response | 44.507 (8.4013) | 56.467 (9.6924)
Statistical Analysis 1: Comparison: Test Platelets Collected and Stored in InterSol vs Control Platelets Collected and Stored in Plasma; The null hypothesis is that HSR's mean difference, Test - 0.8 * Control, is less than or equal to 0, and the alternative is that the mean difference is greater than 0; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; Mean Difference (Final Values) = -0.667, 97.5% CI 1-sided [lower limit -2.499], Standard Deviation 6.7882 — Estimated from an ANCOVA with effects of treatment and subject nested within sequence

6. Secondary Outcome: Platelet Morphology
Description: Quantifies (via phase-contrast light microscopy) the morphological changes of platelets coincident with the full range of platelet activation profile (Units: Kunicki score; Range is 0 to 400). Higher values represent healthier platelets.
Time Frame: Day 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Test Platelets Collected and Stored in InterSol | Control Platelets Collected and Stored in Plasma
Number analyzed (Participants) | 60 | 60
scores on a scale | 293.1 (31.76) | 308.7 (33.30)
Statistical Analysis 1: Comparison: Test Platelets Collected and Stored in InterSol vs Control Platelets Collected and Stored in Plasma; The null hypothesis is that Morphology's mean difference, Test - 0.8 * Control, is less than or equal to 0, and the alternative is that the mean difference is greater than 0; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; Mean Difference (Final Values) = 46.1, 97.5% CI 1-sided [lower limit 40.020], Standard Deviation 23.056 — Estimated from an ANCOVA with effects of treatment and subject nested within sequence

7. Secondary Outcome: Percent of Platelets Activated as Measured by P-selectin
Description: as for outcome 3
Time Frame: Day 7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent of Platelets Activated
Arm/Group | Test Platelets Collected and Stored in InterSol | Control Platelets Collected and Stored in Plasma
Number analyzed (Participants) | 60 | 60
Percent of Platelets Activated | 29.392 (8.0418) | 14.232 (6.4316)
Statistical Analysis 1: Comparison: Test Platelets Collected and Stored in InterSol vs Control Platelets Collected and Stored in Plasma; The null hypothesis is that P-selection's mean difference, Test - 1.25 * Control, is greater or equal to 0, and the alternative is that the mean difference is less than 0; Test type: Non-Inferiority — Lower value is considered to indicate better platelet quality. If the 97.5% upper limit of the confidence interval is less than 0, the null hypothesis will be rejected in favor of the alternative suggesting the Test product is not inferior to the Control product; Mean Difference (Final Values) = 12.314, 97.5% CI 1-sided [upper limit 13.981], Standard Deviation 6.0422 — Estimated from an ANCOVA with effects of treatment and subject nested within sequence

8. Secondary Outcome: Percent of Extent of Shape Change
Description: Measures the proportion of platelets that have a discoid morphology (Units: %). Higher value is considered to indicate better platelet quality. Higher value is considered to indicate better platelet quality.
Time Frame: Day 7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: % of extent of shape change
Arm/Group | Test Platelets Collected and Stored in InterSol | Control Platelets Collected and Stored in Plasma
Number analyzed (Participants) | 60 | 60
% of extent of shape change | 19.328 (6.1433) | 27.962 (5.4495)
Statistical Analysis 1: Comparison: Test Platelets Collected and Stored in InterSol vs Control Platelets Collected and Stored in Plasma; [analysis description as in outcome 4, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; Mean Difference (Final Values) = -3.042, 97.5% CI 1-sided [lower limit -4.407], Standard Deviation 5.4220 — Estimated from an ANCOVA with effects of treatment and subject nested within sequence

9. Secondary Outcome: Percent of Platelets Exhibiting Hypotonic Shock Response
Description: as for outcome 5
Time Frame: Day 7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: % of hypotonic shock response
Arm/Group | Test Platelets Collected and Stored in InterSol | Control Platelets Collected and Stored in Plasma
Number analyzed (Participants) | 60 | 60
% of hypotonic shock response | 37.038 (7.4719) | 49.284 (11.4719)
Statistical Analysis 1: Comparison: Test Platelets Collected and Stored in InterSol vs Control Platelets Collected and Stored in Plasma; [analysis description as in outcome 5, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; Mean Difference (Final Values) = -2.389, 97.5% CI 1-sided [lower limit -4.915], Standard Deviation 9.0544 — Estimated from an ANCOVA with effects of treatment and subject nested within sequence

10. Secondary Outcome: Platelet Morphology
Description: as for outcome 6
Time Frame: Day 7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Test Platelets Collected and Stored in InterSol | Control Platelets Collected and Stored in Plasma
Number analyzed (Participants) | 60 | 60
score on a scale | 269.7 (31.26) | 282.5 (34.79)
Statistical Analysis 1: Comparison: Test Platelets Collected and Stored in InterSol vs Control Platelets Collected and Stored in Plasma; [analysis description as in outcome 6, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; Mean Difference (Final Values) = 43.8, 97.5% CI 1-sided [lower limit 36.821], Standard Deviation 26.05 — Estimated from an ANCOVA with effects of treatment and subject nested within sequence

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events were reported for any participant that underwent any study related apheresis procedure. Only adverse events that occured during the apheresis procedure and until discharge were reported.
Arm/Group | Test Platelets Collected and Stored in InterSol | Control Platelets Collected and Stored in Plasma
All-Cause Mortality (participants affected / at risk) | 0/82 | 0/77
Serious Adverse Events (participants affected / at risk) | 0/82 | 0/77
Other Adverse Events (participants affected / at risk) | 9/82 | 2/77
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test Platelets Collected and Stored in InterSol (N=82) | Control Platelets Collected and Stored in Plasma (N=77)
Injection site extravasation (General disorders) | 7 (7) | 0 (0)
Paraesthesia oral (Nervous system disorders) | 2 (2) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor retains the right to review and comment on any public disclosure of study results. If no response is received within 30 days,the Principal Investigator may presume that the submission for publication may proceed without delay. If the Sponsor asks to defer publication, Study Site shall not publish, or otherwise disclose to any third party, any of the information contained in the publication or presentation until such time as permission is granted from the Sponsor.